CLINICAL TRIAL: NCT02271165
Title: Subcutaneous Immunoglobulin (Hizentra) in Patients With Dermatomyositis: A Proof of Concept Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, marinos dalakas, Professor of Neurology, Thomas Jefferson University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13P.192
Record Dates: First submitted 2014-10-15; First posted 2014-10-22 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — Immunoglobulins; Hizentra; Fluid Therapy

ARMS (2):
- IVIg naive (Active Comparator): Patients naïve to IVIg who have active disease responding to corticosteroids or are corticosteroid-dependent, will be also included. Before these patients enter the study, they will receive 3 monthly infusions of IVIg starting with the standard dose of 2gram/kg/month and followed with monthly maintenance of 1 or 2gram/kg according to their response.
  Interventions: Drug: Immunoglobulin (Hizentra)
- non-IVIg naive (Active Comparator): Participants already on IVIg will be observed for 12 weeks under their existing IVIg regimen and will undergo measurements of their muscle strength, skin changes, assessments of their daily activities and quality of life (QoL) every 4 weeks at scheduled visits for monthly maintenance IVIg infusions (weeks 0,4,8,12).
  Interventions: Drug: Immunoglobulin (Hizentra)

INTERVENTIONS:
Drug: Immunoglobulin (Hizentra)
  Other Names: Immunoglobulin subcutaneous (human) 20% liquid, Hizentra

SUMMARY:
The purpose of the study is to evaluate the effectiveness and safety of human immunoglobulin SCIg in the form of Hizentra (Immune globulin Subcutaneous) in patients with Dermatomyositis. Hizentra provides effective protection against infection by maintaining a steady and normal level of immunoglobulin in the body) in patients with primary immunodeficiency. At present, patients with steroid resistant dermatomyositis can only be treated with IVIg (The healthy antibodies in IVIG can block the damaging antibodies that attack muscle and skin in dermatomyositis) treatment. An evaluation can then be made to see if SCIg is a suitable replacement and exerts immunomodulatory effect on complement antibodies.

ELIGIBILITY:
Inclusion Criteria:

1. Men or woman aged >18 years
2. Diagnosis of DM based on standard criteria
3. Receiving the equivalent of at least 0.4 g/kg IVIg every 4 weeks (IVIg group only)
4. Established response to IVIg or dependence on IVIg to maintain status established either by symptomatic worsening of condition at the end of the inter-dose interval for both groups or by worsening after reduction of the dose within the previous 12 months (IVIg group only)
5. IVIg regimen stable for 12 weeks while on IVIg (minor changes are permitted provided that the dose change is 15% or less) (IVIg group only)
6. Stable dosing with steroids and/or other immunosuppressives for 12 weeks with no changes schedule or intended.

Exclusion Criteria:

1. Pregnancy, planned pregnancy, breast feeding or unwillingness to practice contraception
2. Severe concurrent medical conditions which would prevent treatment or assessment, including significant hematological, renal or liver dysfunction or malignancies
3. Initiation or immunomodulatory treatment other than IVIg in the past 24 weeks or modification of immunomodulatory treatment other than IVIg in the past 12 weeks.
4. Participation in trial of an investigational medicinal product in the past 12 weeks
5. Presence of skin infection unrelated to dermatomyositis, severe skin involvement

Presence of any other medical condition, which in the opinion of the investigator might interfere with performance or interpretation of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-11; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a change in strength (based on MRC sumscores) from baseline (enrollment) to the mean change at weeks 16, 20, 24 and 28. | The primary outcome is a change in strength (based on MRC sumscores) from baseline (enrollment) to the mean change at weeks 16, 20, 24 and 28.
  The primary outcome is a change in strength (based on MRC sumscores) from baseline (enrollment) to the mean change at weeks 16, 20, 24 and 28.

SECONDARY OUTCOMES:
The main secondary outcome is the preference of the participant for SCIg compared with IVIg | The main secondary outcome is the preference of the participant for SCIg compared with IVIg
  Secondary outcome measures will be a) patient preference, based on the number of participants who prefer SCIg to IVIg (a home-made questionnaire will be utilized to capture preference in the most unbiased way; b) average change in Quality of life scores between week 12 and 28; c) effect on the complement consumption in serum; d) Immunological parameters on the repeated skin biopsies; and e) adverse events as reported at each visit. Accordingly, information will be obtained on the superiority of SCIg vs. IVIg

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States